CLINICAL TRIAL: NCT01109225
Title: Multiparametric Study of Cardiac Remodeling After Myocardial Infarction Revascularized in Acute Phase : Relation With the Serum Concentrations in Aldosterone
Brief Title: Relation Between Aldosterone and Cardiac Remodeling After Myocardial Infarction
Acronym: REMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009-A00537-50
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Myocardial Infarction
Keywords: aldosterone; myocardial infarction; cardiac remodeling
MeSH Terms: conditions — Myocardial Infarction | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Myocardial infarction (Experimental): All patients. Patients hospitalized for a first myocardial infarction with known shift of the segment ST revascularized in acute phase by primary angioplasty and dated less than 4 days.
  Intervention:
  * blood sample
  * MRI
  * echocardiography
  * urine sample
  * pulmonary echography
  * vascular check
  * renal echography
  Interventions: Biological: blood sample; Procedure: MRI; Procedure: echocardiography; Biological: urine sample; Procedure: pulmonary echography; Procedure: vascular check; Procedure: renal echography

INTERVENTIONS:
Biological: blood sample
Procedure: MRI
Procedure: echocardiography
Biological: urine sample
Procedure: pulmonary echography
Procedure: vascular check
Procedure: renal echography

SUMMARY:
This study aims to determine whether aldosterone blood levels are predictive of cardiac remodeling at 6 months following myocardial infarction with ST elevation (STEMI), independently of conventional predictive factors (size of myocardial infarction, age, hypertension, etc.) in revascularized patients during the acute phase of MI.

DETAILED DESCRIPTION:
After myocardial infarction, the evolution toward cardiac failure is generally linked to a progressive worsening of cardiac dysfunction and remodeling. Cardiac remodeling is largely the consequence of myocardial injury due to myocardial infarction, although other parameters including age, arterial hypertension, etc. may also represent important predictors. Aldosterone blood levels measured within the first hours of admission for myocardial infarction is associated with increased rates of adverse outcomes. Aldosterone acts on wound healing and fibrosis processes in the myocardium as well as on systemic volemia.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman hospitalized for a first myocardial infarction with known shift of the segment ST revascularized in acute phase by primary angioplasty and dated less than 4 days
* Patient presenting a stable clinical state
* Patient presenting a regular sinusal cardiac rhythm
* Patient having an age ≥ 18 years

Exclusion Criteria:

* Counter-indication with examination MRI
* Severe claustrophobia
* Antecedent of over-sensitiveness to gadolinium salts
* Nonischaemic Cardiopathy
* Cardiac surgery planed in the 6 months
* Women into old to procreate without effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2010-04-27 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
Cardiac remodeling within 6 months of myocardial infarction as defined as the change in left ventricle volumes (increase of more than 20 % of the diastolic volume of the left ventricle) | from initial assessment to 6 months

SECONDARY OUTCOMES:
Vascular and cardiac parameters measured during the initial assesment and at 6 months (both functional and structural - by echocardiography or MRI) | from initial assessment to 6 months
Long-term cardiac remodeling measured by echocardiography at 3 to 9 years of initial enrollment | at 3 to 9 years of initial enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GIRERD, Doctor, Principal Investigator — Centre d'Investigation Clinique Plurithématique 1433/INSERM/CHRU de Nancy
Locations (1):
- Nancy Brabois university hospital, Vandœuvre-lès-Nancy, Meurthe Et Moselle, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Monzo L, Huttin O, Ferreira JP, Lamiral Z, Bozec E, Beaumont M, Micard E, Baudry G, Marie PY, Eschalier R, Rossignol P, Zannad F, Girerd N. Role of aldosterone in mid- and long-term left ventricular remodelling after acute myocardial infarction: The REMI study. Eur J Heart Fail. 2023 Oct;25(10):1742-1752. doi: 10.1002/ejhf.2986. Epub 2023 Aug 24. PMID 37530453
- [Derived] Huttin O, Mandry D, Eschalier R, Zhang L, Micard E, Odille F, Beaumont M, Fay R, Felblinger J, Camenzind E, Zannad F, Girerd N, Marie PY. Cardiac remodeling following reperfused acute myocardial infarction is linked to the concomitant evolution of vascular function as assessed by cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2017 Jan 4;19(1):2. doi: 10.1186/s12968-016-0314-6. PMID 28063459
- [Derived] Huttin O, Marie PY, Benichou M, Bozec E, Lemoine S, Mandry D, Juilliere Y, Sadoul N, Micard E, Duarte K, Beaumont M, Rossignol P, Girerd N, Selton-Suty C. Temporal deformation pattern in acute and late phases of ST-elevation myocardial infarction: incremental value of longitudinal post-systolic strain to assess myocardial viability. Clin Res Cardiol. 2016 Oct;105(10):815-26. doi: 10.1007/s00392-016-0989-6. Epub 2016 Apr 23. PMID 27108156
- [Derived] Huttin O, Petit MA, Bozec E, Eschalier R, Juilliere Y, Moulin F, Lemoine S, Selton-Suty C, Sadoul N, Mandry D, Beaumont M, Felblinger J, Girerd N, Marie PY. Assessment of Left Ventricular Ejection Fraction Calculation on Long-axis Views From Cardiac Magnetic Resonance Imaging in Patients With Acute Myocardial Infarction. Medicine (Baltimore). 2015 Oct;94(43):e1856. doi: 10.1097/MD.0000000000001856. PMID 26512596
- [Derived] Lemarie J, Huttin O, Girerd N, Mandry D, Juilliere Y, Moulin F, Lemoine S, Beaumont M, Marie PY, Selton-Suty C. Usefulness of Speckle-Tracking Imaging for Right Ventricular Assessment after Acute Myocardial Infarction: A Magnetic Resonance Imaging/Echocardiographic Comparison within the Relation between Aldosterone and Cardiac Remodeling after Myocardial Infarction Study. J Am Soc Echocardiogr. 2015 Jul;28(7):818-27.e4. doi: 10.1016/j.echo.2015.02.019. Epub 2015 Mar 31. PMID 25840640
- [Derived] Huttin O, Lemarie J, Di Meglio M, Girerd N, Mandry D, Moulin F, Lemoine S, Juilliere Y, Felblinger J, Marie PY, Selton-Suty C. Assessment of right ventricular functional recovery after acute myocardial infarction by 2D speckle-tracking echocardiography. Int J Cardiovasc Imaging. 2015 Mar;31(3):537-45. doi: 10.1007/s10554-014-0585-7. Epub 2015 Jan 6. PMID 25559651